CLINICAL TRIAL: NCT00397020
Title: A Single-Blind, Randomized, Naturalistic Pilot Study, Comparison of Divalproex ER and Quetiapine for Adults With Acute Mania or Mixed Episodes
Brief Title: Naturalistic Study, Comparison of Divalproex Extended Release (ER) and Quetiapine for Adults With Acute Mania or Mixed Episodes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, David Feifel, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bipolar Mania
Record Dates: First submitted 2006-11-06; First posted 2006-11-08 (Estimated); Results first posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-08

CONDITIONS: Bipolar Disorder
Keywords: quetiapine; divalproex
MeSH Terms: conditions — Bipolar Disorder | interventions — Valproic Acid; Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Divalproex ER (Experimental): Divalproex ER
  Interventions: Drug: divalproex ER
- 2 Quetiapine Fumarate (Active Comparator): quetiapine fumarate
  Interventions: Drug: quetiapine

INTERVENTIONS:
Drug: divalproex ER — Dose: 30mg per kg, rounded to nearest 500mg, dosed PO QHS. Adjustments made through trial to obtain serum valproic acid levels of 85-125 mcg/ml
  Other Names: Depakote ER
  Arms: 1 Divalproex ER
Drug: quetiapine — Dose: 200mg PO QHS, titrated up to therapeutic dose of 600-800mg.
  Other Names: Seroquel
  Arms: 2 Quetiapine Fumarate

SUMMARY:
The primary objective of this study is to compare the efficacy and tolerability of quetiapine versus divalproex extended-release administered in a rapid oral loading fashion in the treatment of acute episodes of mania or mixed mania in bipolar disorder. Three hypotheses will be tested:

Hypothesis 1: treatment ( 3 weeks) of divalproex extended-release is similar to quetiapine in the symptomatic control of mania or mixed mania

Hypothesis 2: divalproex extended-release orally loaded may produce significant improvements in symptoms of mania sooner than quetiapine

Hypothesis 3: divalproex extended-release may produce significantly less sedation

DETAILED DESCRIPTION:
This will be a rater-blinded, head-to-head comparison (no placebo) of divalproex ER and quetiapine in patients with symptoms of an active manic or mixed mania (symptoms of mania and depression). Forty subjects are expected to be enrolled. After screening for eligibility, eligible subjects will be randomized while hospitalized in a 1:1 ratio into 2 treatment groups: divalproex ER or quetiapine. Depakote® ER will be given orally at 30 mg/kg day initially taken at night and rounded up to nearest 500 mg dose with adjustments made through the trial as needed to obtain serum valproic acid levels of 85-125 mcg/ml. Quetiapine will be given orally at an initial dose of 200mg/day on Day 1, and titrate up to 800 mg/day. The duration of the study will be 21 days from baseline and the total number of visits including screening is five. Patients will be released from the hospital once stable and visits for the study will then take place on an outpatient basis.

ELIGIBILITY:
Inclusion Criteria:

For inclusion, patients must fulfill all of the following criteria at enrollment:

1. Provide written informed consent before initiation of any study-related procedures
2. A diagnosis of Bipolar I Disorder, Most Recent Episode Manic (296.4x), or Bipolar I Disorder, Most Recent Episode Mixed (296.5x), with or without psychotic features, as defined by Diagnostic and Statistical Manual of Mental Disorders- Fourth Edition (DSMIV)
3. Male or female, at least 18 years old
4. YMRS score equal to or greater than 17 and a CGI of 4 (moderate) or greater.
5. Female patients of childbearing potential must be using a reliable method of contraception. Reliable methods of contraception include hormonal contraceptives (e.g., oral contraceptive or long-term injectable or implantable hormonal contraceptive), double-barrier methods (e.g., condom and diaphragm, condom and foam, condom and sponge), intrauterine devices, and tubal ligation.

Exclusion Criteria:

1. Known intolerance or lack of response to quetiapine fumarate or Divalproex ER as judged by the investigator.
2. Unwilling or not able to provide informed consent
3. Positive urine toxicology result on screening for cocaine, phencyclidine (PCP), opiates or amphetamines that confirms the current manic/mixed episode is better accounted by a substance intoxication or withdrawal as judged by PI.
4. History of schizophrenia or schizoaffective disorder
5. Treatment with a depot antipsychotic within 1 treatment cycle
6. Unstable medical condition including hepatic, renal, gastroenterologic, neurologic, immunologic, or hematologic diseases that is deemed by the principle investigator to likely to result in hospitalization in 6 months or death within one year
7. A female subject who is pregnant or lactating
8. Lorazepam will be provided for agitation and insomnia as needed for rescue only. Not to exceed 6 mg in the first 7 days; Not to exceed 4 mg for the next 3 days and note to exceed 2 mg/day for the remainder of the study. Those that require a greater amount of Lorazepam will be excluded.
9. Hospitalized for more than 1 week for current episode at the screen
10. Substance or alcohol dependence at enrollment and within the three months prior to enrollment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by DSM-IV criteria.
11. Known diagnosis of dementia or MCI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Feifel, MD, PhD, Principal Investigator — UCSD
Locations (1):
- UCSD Medical Center, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1 Divalproex ER | 2 Quetiapine Fumarate
Started | 14 | 16
Completed | 13 | 15
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Divalproex ER | 2 Quetiapine Fumarate | Total
Number analyzed (Participants) | 13 | 15 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 15 | 28
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 42.4 [19 to 64] | 36.9 [19 to 64] | 39.65 [19 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  United States | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Primary Measure: Young Mania Rating Scale (YMRS) Primary Endpoint: Day 7
Description: Minimum: 0 Maximum: 60 Higher scores indicate worse outcome
Time Frame: Day 7
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | 1 Divalproex ER | 2 Quetiapine Fumarate
Number analyzed (Participants) | 10 | 15
units on a scale | 14.8 (2.1) | 13.9 (1.9)

2. Secondary Outcome: Young Mania Rating Scale (YMRS) Secondary Endpoints
Time Frame: weekly - Day 3, 14, 21
Reporting Status: Not Posted

3. Secondary Outcome: Clinical Global Impression: Severity (CGI:S)
Time Frame: each visit
Reporting Status: Not Posted

4. Secondary Outcome: Clinical Global Impression: Improvement (CGI:I)
Time Frame: each week/visit
Reporting Status: Not Posted

5. Secondary Outcome: Readiness to Discharge Questionnaire (RDQ)
Time Frame: each week/visit in the hospital
Reporting Status: Not Posted

6. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Time Frame: each week/visit
Reporting Status: Not Posted

7. Secondary Outcome: Behavioral Activity Rating Scale (BARS)
Time Frame: each week/visit
Reporting Status: Not Posted

8. Secondary Outcome: Extrapyramidal Symptoms Rating Scale (ESRS)
Time Frame: each week/visit
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | 1 Divalproex ER | 2 Quetiapine Fumarate
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/15
Other Adverse Events (participants affected / at risk) | 1/13 | 5/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Divalproex ER (N=13) | 2 Quetiapine Fumarate (N=15)
Neurological (fainting, dizziness, headaches) (Nervous system disorders) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes